CLINICAL TRIAL: NCT04751955
Title: A Phase lb/ll, Multicenter, Open Label, Single Arm Study to Assess the Safety and Efficacy of the Anti-VEGFR2 Monoclonal Antibody Olinvacimab and the Capecitabine in Patients With mCRC Who Failed Two Prior Chemotherapies
Brief Title: A Phase lb/ll, Open Label, Single Arm Study With Olinvacimab and Capecitabine in mCRC Patients (OLCAP)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This clinical trial was not finally approved by the Korea FDA.
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, SoohyeonLee, Assistant Professor, Korean Cancer Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLCAP
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olinvacimab plus Capecitabine (Experimental): A single arm study with Olinvacimab plus Capecitabine
  Interventions: Drug: Olinvacimab added to Capecitabine

INTERVENTIONS:
Drug: Olinvacimab added to Capecitabine — Olinvacimab: IV weekly administration In phase lb, 12mg/kg and 16mg/kg weekly IV will be tested. In phase ll, the RP2D in phase lb will be used. Capecitabine: fixed dose as an oral administration, 1250mg/m2 BID on day 1 to 14 followed by 7 days off
  Other Names: Capecitabine

SUMMARY:
The aim on this study is to assess the safety and efficacy of the anti-VEGFR2 monoclonal antibody olinvacimab and the capecitabine in patients with metastatic colorectal carcinoma who failed two prior chemotherapies

DETAILED DESCRIPTION:
This is a phase lb/ll, multicenter, open label, single arm study to assess efficacy and safety of the anti-VEGFR2 monoclonal antibody olinvacimab and capecitabine in patients with metastatic colorectal cancer who failed two prior standard chemotherapies.

The primary objective of phase lb is to determine maximal tolerated dose (MTD) and recommended phase ll dose (RP2D) of olinvacimab in combination with capecitabine. the primary objective of phase ll is to assess the efficacy of olinvacimab plus capecitabine as a salvage regimen in metastatic colorectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Phase Ib: Subjects with a histologically-confirmed, advanced/recurrent colorectal cancer who have progressed on two prior standard chemotherapies Phase II: Histologically or cytologically confirmed colorectal cancer patient who had progressed on, were intolerant of, or were inappropriate for the treatment with fluoropyrimidine, oxaliplatin, irinotecan and targeted agents (If the subject received adjuvant chemotherapy after curative surgery and lymph node dissection for colorectal cancer, the adjuvant chemotherapy is considered to be the first-line palliative chemotherapy if the disease recurred during adjuvant chemotherapy or within 6 months after the completion of adjuvant chemotherapy.)
2. Permit previous 2 lines of anti-VEGF blockades
3. Patient has evaluable disease as per RECIST 1.1. (Measurable lesions are not mandatory for study inclusion.)
4. Age ≥ 19 years old of male and female
5. ECOG performance status (PS) 0-1
6. Adequate bone marrow and organ function as defined by the following laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
   * Platelet ≥ 75 x 109/L
   * Serum creatinine ≤ ULN (upper limit of normal) x 1.5 or serum creatinine clearance > 30 mL/min
   * Total bilirubin: ≤ 2.0 × ULN, Subjects with a bile duct obstruction will be eligible if they meet the criteria after appropriate bile drainage
   * Phase Ib: Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 3 x ULN (regardless of liver metastases)
   * Phase II: AST and ALT ≤ 3 x ULN if liver metastases are absent, or AST and ALT ≤ 5 x ULN if liver metastases are present.
7. Adequate cardiac function: QTc ≤480 msec; if QTc exceeds 480 msec, subjects can be enrolled if the average QTc value is less than 480 msec by measuring 3 times consecutively in total.
8. The subject is able to swallow and retain oral medication
9. Serum β-HCG test negative within 14 days before the first administration of the study treatment (women of childbearing potential only).
10. Requirement for contraception must be observed by the subject.
11. Life expectancy of at least 3 months
12. Subject has signed the Informed Consent Form (ICF) prior to any screening procedures being performed.

Exclusion Criteria:

1. Patient has a known or suspicious hypersensitivity to fluoropyrimidines.
2. Any cytotoxic chemotherapy from a previous treatment regimen within 14 days. If the subject received an investigational drug from another clinical trial, the subject can be enrolled after 2 weeks of last administration and more than 5 x half-life of the investigational drug. If monoclonal antibody therapy including anti VEGF agent was given, the subject can be enrolled after four weeks after the last does.
3. Patients with complete or partial dihydropyrimidine dehydrogenase deficiency.
4. Serious uncontrolled intercurrent infections
5. Serious intercurrent medical or psychiatric illness, including active cardiac disease

   * Acute coronary syndrome within the 6 months prior to the initiation of study drug (including myocardial infarction or unstable angina, Coronary Artery Bypass Graft surgery, percutaneous coronary intervention and stenting)
   * Heart failure ≥ grade 2 by New York Heart Association (NYHA) functional classification or that requires treatment
   * Ejection fraction (EF) <50% on multi-gated acquisition (MUGA) scan or echocardiography examination. MUGA scan or echocardiography is not required as a screening test if there is no current suspicious symptom and past history of heart failure.
   * Persistent uncontrolled hypertension as defined by: systolic >180 mmHg or diastolic >100 mmHg despite medical treatment. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
   * Current or past history of clinically significant cardiac arrhythmia, atrial fibrillation, and/or conduction abnormality (e.g. congenital long QT syndrome, complete AV block)
   * Any risk factors that prolong QTc or increase the probability of arrhythmia, including medication (e.g. heart failure, hypokalemia, congenital long QT syndrome, history of Torsades de Pointes)
6. Active central nervous system (CNS) lesions (i.e., those with radiologically unstable or symptomatic brain lesions). For those who receive radiation or surgical treatment, the subject can be enrolled if the subject is maintained without steroid therapy and the evidence of CNS disease progression for more than 4 weeks. However, patients with leptomeningeal metastases are excluded.
7. History of other primary cancer. Exceptions are as follows:

   * Adequately treated non-melanoma skin cancer (basal cell or squamous cell carcinoma), curatively treated in situ cancer of the cervix or stage I bladder cancer, completely resected thyroid cancer without distant metastasis in which all treatment has been completed (Appropriate wound healing is required prior to clinical trial enrollment)
   * Other curatively treated solid tumors except for gastric cancer with no evidence of disease recurrence at least 36 months before participating in this trial
8. Patient has not recovered to ≤ grade 1 (except alopecia) from related adverse effects of any prior antineoplastic therapy.
9. Radiotherapy with a wide field (more than 30% of the bone marrow) of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
10. Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from adverse effects of such procedure.
11. Patient has a known positive serology for human immunodeficiency virus (HIV), active Hepatitis B, and/or active Hepatitis C infection. Hepatitis B carriers may be enrolled if prophylactic use of an antiviral agent with minimal interaction with CYP3A4 is administered to inhibit HBV activation (e.g., entecavir, adefovir)
12. Concomitant medication of strong or moderate inducers or inhibitors of CYP3A4 before the first dose of study treatment (In this case, if the drug is stopped for more than 1 week and changed to another drug that does not affect CYP3A4, then the subject can be enrolled.)
13. People who are taking BCRP inhibitors, allopurinol, soribudin, brivudine or within 4 weeks of stopping, and taking tegafur/gimeracil/oteracil or within 7 days of stopping
14. History of allogeneic bone marrow transplantation or organ transplantation
15. As judged by the Investigator, all other symptoms and associated disease for which the investigator determined that participation in this study is contraindicated (e.g. Infection/inflammation; severe liver dysfunction; bilateral diffuse interstitial lung disease; uncontrolled renal disease; unstable heart and lung disease; hemorrhagic disease; intestinal obstruction; unable to swallow oral pills; social and psychological problems, etc.)
16. Medical, psychiatric, cognitive, or other conditions that may interfere with the ability of the subject to understand the subject information, provide the informed consent, follow the protocol process, or complete the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) | Through phase 1b, up to 6 month
  recommended phase ll dose (RP2D) of olinvacimab in combination with capecitabine
Progression free survival | 3 years
  Progression free survival of olinvacimab plus capecitabinel

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Determination of the ORR will be calculated based on the proportion of patients achieving CR or PR using the RECIST v1.1 as assessed by investigators.
overall survival | 3 years
  overall survival
Disease control rate (DCR) | 2 years
  DCR will be calculated based on the proportion of patients achieving CR, PR, or who have SD at least 6 weeks after receiving first dose of study treatment.
Duration of response (DOR) | 2 years
  DOR will be calculated from the time of initial response (CR or PR) documentation to the time of progressive disease (PD). If a subject who had CR or PR dies without the evidence of disease progression, the case will be censored at the time point of death when analyzing DOR
Time to response (TTR) | 2 years
  Time to response (TTR) will be calculated from the first dose of study drug to the time point of initial response (CR or PR).
Toxicity by CTCAE v5.0 | 3 years
  Safety assessments should be conducted for all subjects who received olinvacimab plus capecitabine at least once. Adverse events will be graded according to CTCAE v5.0.
Quality of life by FACT-C v4.0 | 2 years
  Quality of life as measured by FACT-C v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Soohyeon Lee, MD, PhD, Principal Investigator — Korea Cancer Study Group

IPD SHARING:
Plan to Share IPD: No